CLINICAL TRIAL: NCT06701994
Title: Efficacy of an Innovative Kinesiotaping Bandage Compared to Traditional Tape in Stabilising Ankle Inversion and Plantar Flexion in Triathletes: A Triple-Blind Experimental Study
Brief Title: Efficacy of an Innovative Kinesiotaping Bandage Compared to Traditional Tape in Stabilising Ankle Inversion and Plantar Flexion in Triathletes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Hernandez-Lucas, Phd, University of Vigo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Vendaje Ogando
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Athletes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesiotaping Bandage Group (Experimental): A bandage using kinesiotape will be applied to the participant's ankle directly on the skin and covered with an opaque stocking.
  Interventions: Behavioral: Innovative Kinesiotaping Bandage Group
- Traditional Tape Bandage Group (Active Comparator): A bandage will be applied to the participant's ankle using kinesiotape directly on the skin and covered with an opaque stocking.
  Interventions: Behavioral: Traditional Tape Bandage Group
- Placebo Group (Placebo Comparator): An opaque stocking is placed on the participant's ankle.
  Interventions: Behavioral: Placebo Bandage Group

INTERVENTIONS:
Behavioral: Innovative Kinesiotaping Bandage Group — This group will receive an innovative kinesiotaping bandage developed specifically for this study. The kinesiotape will be applied directly to the skin on the ankle, combining water resistance with restrictive properties to stabilise the joint while maintaining flexibility. Unlike traditional tape, the kinesiotape is designed to perform well in aquatic conditions, making it suitable for triathlon demands. It provides joint support while allowing a greater range of motion, aiming to enhance performance across all phases of the sport. To maintain blinding, the bandage will also be covered with an opaque stocking.
  Arms: Kinesiotaping Bandage Group
Behavioral: Traditional Tape Bandage Group — Participants in this group will receive a traditional ankle bandage using functional tape. The bandage is applied directly to the skin and is designed to restrict ankle inversion and plantar flexion, providing stability to prevent recurrent injuries. Traditional tape bandages are widely used in sports due to their effective joint stabilisation. However, they have significant limitations in aquatic environments as they lack water resistance, which makes them less effective during the swimming phase of triathlons. The bandage will be covered with an opaque stocking to ensure blinding, preventing participants or evaluators from identifying the type of intervention.
  Arms: Traditional Tape Bandage Group
Behavioral: Placebo Bandage Group — Participants in this group will receive a placebo bandage consisting of a simple gauze wrap applied directly to the ankle. The gauze lacks stabilising or therapeutic properties and is used as a control to account for potential placebo effects. Although it mimics the application process of the other bandages, it does not provide functional or structural support to the ankle joint. An opaque stocking will cover the gauze to ensure that neither participants nor evaluators can distinguish the placebo bandage from the others, maintaining the integrity of the blinding process.
  Arms: Placebo Group

SUMMARY:
Efficacy of an Innovative Kinesiotaping Bandage Compared to Traditional Tape in Stabilising Ankle Inversion and Plantar Flexion in Triathletes: A Triple-Blind Experimental Study.

Background and Purpose:

Lateral ankle sprains are a common injury among triathletes, impacting their performance and recovery time. Although traditional functional tape is effective in stabilising the ankle joint, it has limitations in aquatic sports due to its lack of water resistance. This study will evaluate the efficacy of an innovative kinesiotaping (KT) bandage, designed to combine water resistance with the restrictive properties of traditional tape. The primary objective will be to determine which type of bandage is more effective in stabilising ankle inversion and plantar flexion in triathletes.

Study Design:

This will be a triple-blind experimental study involving 20 federated triathletes. Each participant will have three different bandages (traditional tape, innovative KT, and placebo) applied in a randomised order. Goniometric and functional tests will be used to measure the outcomes.

Interventions:

Traditional Tape: Standard restrictive bandage. Innovative KT Bandage: Elastic, water-resistant bandage with additional restrictive properties.

Placebo: Gauze bandage without stabilising properties.

Methods of Evaluation:

Goniometric measurements (flexion, inversion) and functional tests (Star Excursion Balance Test, Hopping Test, Vertical Jump Test) will be conducted. The bandages will be applied and evaluated in a controlled environment, with participants and investigators blinded to the type of bandage.

Expected Outcomes:

It is anticipated that the innovative KT bandage will provide stabilisation comparable to traditional tape for critical ankle movements while overcoming the limitations of tape in aquatic conditions. It is also expected to demonstrate significant advantages in functional tests.

Clinical Relevance:

This study aims to provide evidence for optimising the management of ankle injuries in triathletes, offering a practical and effective solution to maintain athletic performance under demanding conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult men (over 18 years old).
* Federated triathletes.
* No medical conditions or pathologies that could affect the measurements.
* Signed informed consent.

Exclusion Criteria:

* Recent surgeries that compromise ankle function.
* Severe prior ankle injuries (fractures, ligament tears).
* Presence of chronic musculoskeletal diseases.
* Use of ankle support devices during the tests.
* History of severe dermatological allergies or intolerance to the materials used in the bandages.
* Use of supplements or medications that could influence muscular or joint performance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Ankle Goniometry | From enrollment to the end of measurements, approximately one hour
  The ankle's range of motion was evaluated, including dorsiflexion, plantar flexion, eversion, and inversion. Three measurements were taken for each movement, and their mean value was calculated using a GemRed® digital goniometer. The procedure was conducted while ensuring the patient's proper positioning and aligning the instrument with anatomical reference points.

SECONDARY OUTCOMES:
Star Excursion Balance Test | From enrollment to the end of measurements, approximately one hour.
  Dynamic postural control was evaluated through a test in which participants, while maintaining balance on their dominant foot, had to reach the furthest point in each of the eight directions of a star. Distances were measured from the centre of the supporting foot to the tip of the opposite foot. To obtain a general indicator of dynamic balance performance, the average of the distances reached in all directions was calculated.
Hopping Test | From enrollment to the end of measurements, approximately one hour.
  The Hopping Test evaluates dynamic balance and agility on uneven surfaces. Participants perform a hopping sequence over elevated squares tilted at a 15° angle. The task involves completing a course by hopping back and forth across eight marked squares as quickly as possible, maintaining balance and control. The total time required to complete the course is recorded as the performance outcome. This test assesses functional stability and proprioception under challenging conditions.
Vertical Jump Test | From enrollment to the end of measurements, approximately one hour.
  The Vertical Jump Test measures explosive lower-limb strength and power. Participants perform two types of jumps: a countermovement jump and a squat jump from a static position. A force platform records flight time and calculates jump height for each attempt. The test evaluates the participant's ability to generate power in vertical motion, providing insights into muscular performance and functional capacity. Results are analysed to compare performance across conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontevedra, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No